CLINICAL TRIAL: NCT04218500
Title: Comparison of the Effectiveness and Safety Between Moisturizing Cream Containing Niacinamide 4% and Virgin Coconut Oil 30% for Secondary Prevention of Occupational Hand Hermatitis in Intensive Care Unit Nurses: a Double Blind Randomized Clinical Trial
Brief Title: The Effectiveness and Safety of Niacinamide 4% and Virgin Coconut Oil 30% for Secondary Prevention of Occupational Hand Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yenny Rachmawati, Principal investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IndonesiaDV
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-09

CONDITIONS: Contact Dermatitis of Hands
Keywords: Occupational Hand Dermatitis; Moisturizer; Niacinamide; Virgin coconut oil; HECSI; TEWL; SCap

STUDY DESIGN:
Intervention Model Description: There were 46 subjects in the niacinamide 4% arm and 46 subjects in the VCO 30% arm
Who Masked: Participant, Investigator
Masking Description: Both moisturizers have the same physical characteristics, with the same color and odor.
  Randomization was carried out by other than researcher (statistical adviser)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niacinamide 4% (Active Comparator): Niacinamide 4%, applied twice daily for 28 days
  Interventions: Other: Niacinamide 4%
- Virgin coconut oil 30% (Active Comparator): Virgin coconut oil 30%, applied twice daily for 28 days
  Interventions: Other: Virgin Coconut oil 30%

INTERVENTIONS:
Other: Niacinamide 4% — cream moisturizer
  Arms: Niacinamide 4%
Other: Virgin Coconut oil 30% — cream moisturizer
  Arms: Virgin coconut oil 30%

SUMMARY:
Occupational hand dermatitis (OHD) often occurs in intensive care unit (ICU) nurses, especially in individuals who are vulnerable due to irritant exposure e.g. hand rub alcohol and repeated hand washing activities. The use of moisturizer is one of the recommendations for skin care in OHD. Niacinamide which has anti-inflammatory effects and can improve the skin barrier function. Virgin coconut oil (VCO) is rich in lipids and lauric acid, and has an occlusive effect. Until now there are no guidelines and reference types of moisturizers for secondary prevention in DTAK.

DETAILED DESCRIPTION:
The aim of this study is identify the effectiveness and safety between moisturizing cream containing niacinamide 4% and VCO 30% for secondary prevention of occupational hand dermatitis in ICU nurses This study also measured HECSI , TEWL, and SCap before and after treatment

ELIGIBILITY:
Inclusion Criteria:

ICU nurses who:

* Sign the informed consent of the study after receiving explanation before all activity related with this study begin.
* Has Occupation Hand Dermatitis that fulfill the Mathias criteria with dermatitis severity mild to moderate which the score is 1, 2 or 3 corresponding with Investigator Global Assesment (IGA)
* Agree to follow the study protocol

Exclusion Criteria:

* History of allergic or irritate by Niacinamide or VCO or other component in moisturizer
* Receiving medium to high potency of topical Corticosteroid or systemic immunosupresant therapy or history of oral corticosteroid therapy in the last 1 month

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
HECSI | 14 days
  Hand eczema severity index (HECSI) is a score to indicate the severity of hand dermatitis. The range of HECSI score is 0-360. The HECSI score before treatment was expected to be higher than after treatment. Outcome: change of HECSI
HECSI | 28 days
  Hand eczema severity index (HECSI) is a score to indicate the severity of hand dermatitis. The range of HECSI score is 0-360. The HECSI score before treatment was expected to be higher than after treatment. Outcome: change of HECSI
TEWL | 14 days
  Trans Epidermal Waterloss (TEWL) is the primary parameter which measured for the skin barrier function, when the skin barrier is damaged the skin will be disrupted in maintaining water. Passive water diffusion via the Corneal stratum. TEWL is measured in g/h/m2. The TEWL value before treatment was expected to be higher than after treatment. Outcome: change of TEWL
TEWL | 28 days
  Trans Epidermal Waterloss (TEWL) is the primary parameter which measured for the skin barrier function, when the skin barrier is damaged the skin will be disrupted in maintaining water. Passive water diffusion via the Corneal stratum. TEWL is measured in g/h/m2. TEWL value before treatment was expected to be higher than after treatment. Outcome: change of TEWL
SCap | 14 days
  Skin Capasitance (SCap) is a score for skin hidration. SCap can be done with measuring the water level in corneal stratum using non-invasive electric method which measure the capacitance. SCap is measured in Arbitrary Unit (AU). SCap value before treatment was expected to be lower than after treatment. Outcome: change of SCap
SCap | 28 days
  Skin Capasitance (SCap) is a score for skin hidration. SCap can be done with measuring the water level in corneal stratum using non-invasive electric method which measure the capacitance. SCap is measured in Arbitrary Unit (AU). SCap value before treatment was expected to be lower than after treatment. Outcome: change of SCap.

CONTACTS AND LOCATIONS:
Overall Officials: Dermatology and Venereology Departement, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No